CLINICAL TRIAL: NCT03131232
Title: The Aim of This Study is to Investigate the Protective Effect of Empagliflozin on the Cardiovascular System in Diabetes Mellitus Patients
Brief Title: The Effect of Empagliflozin on Glucose Metabolism, Weight, Blood Pressure and Cardiac Function (NT-proBNP) Should be Investigated
Acronym: Empa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-152
Record Dates: First submitted 2017-04-13; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In summary, the registry should provide novel insight into potential mechanisms of cardiovascular risk reduction in patients treated with Empagliflozin with an indication of intensified glucose lowering therapy based on their HbA1c level.

DETAILED DESCRIPTION:
Patients with diabetes exhibit an increased risk for the development of cardiovascular disease with a significantly impaired prognosis compared to patients without diabetes. Recent data from the EMPA-REG Outcome Trial suggest that treatment with the SGLT-2 inhibitor Empagliflozin reduces cardiovascular events, cardiovascular mortality as well as hospitalization for heart failure in patients with type 2 diabetes and pre-existing cardiovascular disease. Empagliflozin leads to reduction of blood glucose by an increased glucose excretion reduces blood pressure and weight. Still, it remains unclear how empagliflozin led to this pronounced reduction of cardiovascular mortality the EMPA-REG OUTCOME trial. Thus, our registry will analyse various biochemical as well as clinical markers in patients with type 2 diabetes and newly initiated treatment with empagliflozin. and an indication for intensification of glucose lowering therapy with empagliflozin. Patients with an indication for an intensified glucose-lowering therapy (HbA1c > 7,5%) will receive 10 mg empagliflozin and we will perform biochemical analyses of blood samples including insulin, glucagon as well as metabolites at baseline as well as after 1 and 6 months. In addition we will assess echocardiographical data.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus II Patients with whom an empagliflozine treatment is to be initiated from a clinical indication

Exclusion Criteria:

* Inability to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: If possible, all patients of the Department MK1 Uniklinik Aachen who are treated with empagliflozine
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of empagliflozine on glucose metabolism | 6 month
  HbA1c in %
The effect of empagliflozine on glucose metabolism | 6 month
  Body weight in kg
The effect of empagliflozine on glucose metabolism | 6 month
  BMI in kg/m²
The effect of empagliflozine on glucose metabolism | 6 month
  blood pressure in mmHg
The effect of empagliflozine on glucose metabolism | 6 month
  NT-pro BNP in pg/ml

SECONDARY OUTCOMES:
Frequency of urinary and urogenital infections | 6 month
  Urinary infection as reported by the patient CRP (Creactive protein) in mg/dl
detection differential regulation of endogenous and exogenous metabolites in addition to circulating proteins by empagliflozin. | 6 month
  perform metabolomic and proteomic profiling of serum samples
Lipid measurements | 6 month
  LDL-C in mg/dl HDL-C in mg/dl TG (triglyceride) in mg/dl
- echocardiographic parameters (if collected) with determination of the systolic and diastolic left ventricular function | 6 month
  LV-EF (left ventricular ejection fraction) in % LV (left ventricular) global strain

CONTACTS AND LOCATIONS:
Overall Officials: Dirk DM Müller Wieland, Scientific Director, Study Director — Coordination Center for Clinical Study

IPD SHARING:
Plan to Share IPD: No